CLINICAL TRIAL: NCT03647384
Title: Efficacy and Safety of Guilingji Capsule in Older Adults With Mild-to-Moderate Cognitive Impairment (Kidney and Marrow Deficiency Pattern)
Brief Title: Guilingji Capsule for Mild-to-moderate Cognitive Impairment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); Beijing Xuanwu Traditional Chinese Medicine Hospital (Unknown); Beijing Hospital (Other Government); Beijing Shijitan Hospital, Capital Medical University (Other); Peking University First Hospital (Other); Huadong Hospital (Other); Longhua Hospital (Other); The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); The Affiliated Hospital of Shandong University of TCM (Unknown); Shanxi Dayi Hospital (Other); Shaanxi Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Li Hao, Study Chair, Xiyuan Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2018XLA039-2
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Cognitive Dysfunction
Keywords: Traditional Chinese medicine; Randomized clinical trial; Mild-to-moderate cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants are randomly and evenly assigned to 2 groups using block randomization.Random numbers are generated by the stratified random method using the SAS statistical software and assigned by an independent statistician at the Good Clinical Practice Institute of Xiyuan Hospital. Drugs are numerically labeled and sequenced according to the random numbers. The drug randomization is conducted by drug supplier. The patients are assigned to the intervention according to the sequence.
  The clinicians, patients and statistician are blind to the patients' grouping assignment and intervention. Database is locked after all data is inputted. The grouping information will be revealed when statistical analyses are conducted. The researchers reveal the second blinding and write the study report finally. Unblinding is allowed only in emergency situation for the patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In this arm, patients take 0.6g of Gulingji capsules, 2 hours before breakfast, served with light salt water once a day. Also an oral take of 19.2mg Ginko Biloba Extract mimetic three times a day. Treatment lasts for 24 weeks.
  Interventions: Drug: Gulingji capsules
- Control (Active Comparator): In this arm, patients take 0.6g of Gulingji mimetic, 2 hours before breakfast, served with light salt water once a day. Also an oral take of 19.2mg Ginko Biloba Extract tablet three times a day. Treatment lasts for 24 weeks.
  Interventions: Drug: Ginko Biloba Extract tablet

INTERVENTIONS:
Drug: Gulingji capsules — Patients take 0.6g of Gulingji capsules, 2 hours before breakfast, served with light salt water once a day. Also an oral take of 19.2mg Ginko Biloba Extract mimetic three times a day. Treatment lasts for 24 weeks.
  Arms: Intervention
Drug: Ginko Biloba Extract tablet — Patients take 0.6g of Gulingji mimetic, 2 hours before breakfast, served with light salt water once a day. Also an oral take of 19.2mg Ginko Biloba Extract tablet three times a day. Treatment lasts for 24 weeks.
  Arms: Control

SUMMARY:
This study is aiming to evaluate the efficacy and safety of Guilingji capsule in older adults with mild-to-moderate cognitive impairment who diagnosed as the kidney and marrow deficiency pattern in TCM. A total of 348 participants are evenly assigned to two arms. In the intervention arm, participants receive Guilingji capsule and Ginko Biloba Extract mimetic in combination, while the other arm will receive Ginko Biloba Extract tablet with Gulingji mimetic.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, positive control, noninferiority clinical trials. Experimental arm (174 cases) take 0.6 g of Gulingji capsules once a day and 19.2 mg of Ginko Biloba Extract mimetic three times a day. Active Comparator arm (174 cases) should take 0.6 g of Gulingji mimetic once a day and 19.2 mg of Ginko Biloba Extract tablet three times a day. The intervention lasted for 24 weeks. Clinical researchers, participants and statisticians are blinded to the treatment assignment throughout the study. Co-primary efficacy endpoints are change from baseline to week 12 and 24 in Mini-Mental State Examination score and Montreal Cognitive Assessment (MoCA) total score.Change from baseline to week 12 and 24 in Clinical Dementia Rating score, Alzheimer's Disease Assessment Scale-Cognitive subscale score, Activities of Daily Living, and Chinese Medicine Symptom Scale scoreare additional endpoints. Prespecified secondary biomarker endpoint is change from baseline in the serum level of acetylcholine and acetylcholinesterase at week 24.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 60 and 85 years old
2. With a disease course ≥ 6 months and confirmed by others
3. Mini-Mental State Examination (MMSE) score between 10 and 26, or MMSE score >26 but Montreal Cognitive Assessment (MoCA) score<26
4. Meeting the diagnostic criteria of mild-to-moderate cognitive impairment
5. Meeting the diagnostic criteria of kidney deficiency pattern in Traditional Chinese medicine
6. Screening visit brain MRI and CT scan consistent with the diagnosis of mild-to-moderate cognitive impairment
7. Adequate visual and auditory abilities to perform all aspects of the cognitive and functional assessments
8. Received a primary and/or a higher education
9. Lives at home with appropriate caregiver capable of accompanying the subject on all clinic visits, or community dwelling with caregiver capable of accompanying the subject on all clinic visits and visiting with the subject approximately 5 times per week for the duration of the study
10. Signed and dated written informed consent. The subject's caregiver must also consent to participate in the study

Exclusion Criteria:

1. Significant neurological disease, other than AD MCI and VaD, that may affect cognition, such as the Parkinson's disease, the Huntington's disease, normal pressure hydrocephalus, brain tumors, progressive supra-nuclear palsy, epilepsy, chronic subdural hematoma and multiple sclerosis, history of severe head trauma with persistent neurological deficits or known abnormal brain structure
2. Thyroid disease, vitamin B12 or folic acid deficiency, severe anemia or malnutrition, serious heart, liver, lung, kidney and other organ diseases that may affect the cognitive function
3. Allergic to Ginkgo products
4. Use of any other medications with the potential to affect cognition
5. Current presence of a clinically important major psychiatric disorder or symptom
6. Alcohol addiction, or long-term use of antipsychotic drugs, or a history of severe head trauma
7. Cannot complete with cognitive function examines.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2018-08-22 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The Change From Baseline in Mini-Mental State Examination (MMSE) Total Score at Week 12 and 24 | Baseline,12th week±3 days, 24th week±3 days
  MMSE is a 30-point questionnaire and contains items assessing orientation, memory, attention and calculation, naming and visuospatial skills of patients.
The Change From Baseline in Montreal Cognitive Assessment (MoCA) Total Score at Week 12 and 24 | Baseline,12th week±3 days, 24th week±3 days
  MoCA is a 30-point questionnaire and evaluates orientation, executive function, language ability, short-term memory, attention and visuospatial ability.

SECONDARY OUTCOMES:
The Change From Baseline in Clinical Dementia Rating (CDR) Total Score at Week 12 and 24 | Baseline,12th week±3 days, 24th week±3 days
  The CDR test is a numeric scale used to quantify the severity of symptoms of dementia. It sums 6 clinical ratings: 1) memory, 2) orientation, 3) judgment and problem solving, 4) involvement in community affairs, 5) home and hobbies, and 6) personal care based on the CDR interview. The CDR includes discussions with the participant and caregiver using a structured format. CDR total score range is 0 (least impairment) to 18 (most impairment); a negative change from baseline indicates an improvement.
The Change From Baseline in the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) Total Score at Week 12 and 24 | Baseline,12th week±3 days, 24th week±3 days
  The ADAS-Cog is a multi-item, objective measure of cognitive function. Analysis of the ADAS-Cog for this study is based upon an 12 item score from the following items 1) word recall task, 2) naming objects and fingers, 3) following commands, 4) constructional praxis, 5) ideational praxis, 6) orientation, 7) word recognition, 8) remembering test instructions, 9) spoken language ability, 10) word finding difficulty in spontaneous speech, 11) comprehension, and 12) attention during the test. The ADAS-Cog ranged from 0 to 75 points, with higher scores indicating a greater degree of impairment. A negative change from baseline indicates a decrease in cognitive impairment.
The Change From Baseline in Activities of Daily Living (ADL) Total Score at Week 12 and 24 | Baseline,12th week±3 days, 24th week±3 days
  The ADL is a test used in healthcare to evaluate the people's daily self care activities.
The Change From Baseline in The Chinese Medicine Symptom Scale (CM-SS) Total Score at Week 12 and 24 | Baseline,12th week±3 days, 24th week±3 days
  The CM-SS is a tool, designed according to the Guiding Principles of Clinical Research on New Drugs of Traditional Chinese Medicine issued in 2002, to evaluate the effects of treatments on Traditional Chinese medicine patterns (here refers to kidney deficiency pattern). Scoring is mainly based on some typical TCM symptoms, such as tongue coating and pulse.
The Change From Baseline in The Serum Level of Acetylcholine and Acetylcholinesterase at Week 24 | Baseline, 24th week±3 days
  Acetylcholine and acetylcholinesterase are potential circulatory biomarkers of cognitive dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Li, Study Chair — Institute of Geriatrics, Xiyuan Hospital, China Academy of Chinese Medical Sciences,
Locations (1):
- Li Hao, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liu NY, Pei H, Liu MX, Liu LT, Fu CG, Li H, Chen KJ. Efficacy and Safety of Guilingji Capsules () for Treating Mild-to-Moderate Cognitive Impairment: Study Protocol for A Randomized, Double-Blind, Positive-Controlled, Multicenter and Noninferiority Trial. Chin J Integr Med. 2020 Aug;26(8):577-582. doi: 10.1007/s11655-020-2723-5. Epub 2020 Aug 5. PMID 32761337